CLINICAL TRIAL: NCT02855853
Title: Study of the Impact of Implicit Motor Training Using a Virtual Reality System and Serious Games on a Tablet Computer in a Rehabilitation Programme in Frail Elderly Subjects
Brief Title: Study of the Impact of Implicit Motor Training in a Rehabilitation Programme in Frail Elderly Subjects
Acronym: MAAMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Other
Other Study IDs: MANCKOUNDIA ANR 2012
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Rehabilitation Frail Elderly Subjects

ARMS (2):
- serious game (Experimental)
  Interventions: Other: serious game et virtual reality
- control (Placebo Comparator)
  Interventions: Other: Nintendo Wii

INTERVENTIONS:
Other: serious game et virtual reality
  Arms: serious game
Other: Nintendo Wii
  Arms: control

SUMMARY:
Even though cognitive-motor performances are impaired in frail elderly subjects compared with healthy elderly subjects, exercising cognitive-motor processes in an implicit manner can improve the carrying out of real actions in everyday life.

No training programme using virtual reality and serious games oriented towards the perception/action system has been tested in frail elderly subjects.

The expected results are:

* In the short term, greater strengthening of motor and cognitive abilities in subjects trained with the virtual reality and serious games, thanks to stimulation through action and through the underlying processes.
* In the long term (+1 and +3 months at the end of the training period) better preservation of motor and cognitive abilities in subjects who took part in the virtual reality and serious games programme.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Who have provided oral consent
* Enrolled in a geriatric rehabilitation programme
* Qualified as cognitively frail, that is to say a MiniMental State Examination (MMSE) score between 15 and 28 and/or for motor abilities, a walking speed less than 0.65 m/s.
* Aged ≥ 65 years
* Able to understand simple instructions

Exclusion Criteria:

Patients:

* Not covered by national health insurance
* With an extremely low cognitive status (MMSE < 15)
* With severely impaired vision and audition (unable to discern any sensory information from the virtual reality system: music, sounds, images)
* Who are unstable when standing
* With an unsteady gait (risk of falling)
* Who cannot walk at least 10 metres
* With an acute non-stabilized cardiovascular disease
* With one or several non-consolidated fractures.
* Under guardianship

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement in performance at the Timed Up and Go (TUG) in the group taking part in the implicit motor training programme compared with a group having conventional motor training. | Change from baseline at Day0 and after 6 weeks of training

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Bourrelier J, Kubicki A, Rouaud O, Crognier L, Mourey F. Mental Rotation as an Indicator of Motor Representation in Patients with Mild Cognitive Impairment. Front Aging Neurosci. 2015 Dec 23;7:238. doi: 10.3389/fnagi.2015.00238. eCollection 2015. PMID 26779010